CLINICAL TRIAL: NCT00838123
Title: Cognitive Functioning Related to Job Tenure Among Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Research Ethics Review Committee, Far Eastern Memorial Hospital
Other Study IDs: FEMH-96-C-044
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this research is to explore which cognitive function would affect the job tenure among people with schizophrenia. The investigators plan to recruit 60 people diagnosed with schizophrenia and divide into two groups, employment and unemployment. The investigators will use several cognitive function tests to collect their cognitive functions and PANSS to evaluate their psychotic symptoms. And then the investigators will compare and analysis the data through statistic software. Finally, the investigators will have the answer about if cognitive functions would affect the job tenure among people with schizophrenia. And the investigators hope that we could get the predict factor of cognitive function to predict the successful employment in future.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia, 18~44y/o

Exclusion Criteria:

* substance abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: schizophrenia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Study Completion 2008-12 (Actual)